CLINICAL TRIAL: NCT05465070
Title: Leg Heat Therapy to Improve Functional Performance in Peripheral Artery Disease
Brief Title: Leg Heat Therapy in Peripheral Artery Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Raghu Motaganahalli, Professor, Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13615; 1R01AG073634-01A1 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Artery Disease
Keywords: heat therapy; peripheral artery disease; walking performance; muscle strength
MeSH Terms: conditions — Peripheral Arterial Disease; Hyperthermia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Heat therapy (Experimental): Patients will be provided with water-circulating trousers, a water heater, and a water tank coupled to a water pump. The heater will be adjusted to warm up the water to 42ºC. Participants will be asked to apply the therapy daily for 90 min while seated or in the supine position.
  Interventions: Device: Leg heat therapy
- Sham Control (Active Comparator): Patients will be provided with water-circulating trousers, a water heater, and a water tank coupled to a water pump. The heater will be adjusted to warm up the water to 33ºC. Participants will be asked to apply the therapy daily for 90 min while seated or in the supine position.
  Interventions: Device: Sham Control

INTERVENTIONS:
Device: Leg heat therapy — A sous vide heating immersion circulator heats up the water inside the water tank to 42ºC. A water pump circulates temperature-regulated water through the trousers.
  Arms: Heat therapy
Device: Sham Control — A sous vide heating immersion circulator heats up the water inside the water tank to 33ºC. A water pump circulates temperature-regulated water through the trousers.
  Arms: Sham Control

SUMMARY:
The goal of this randomized, double-blind, sham-controlled clinical trial is to evaluate the benefits of home-based, leg heat therapy (HT) on lower-extremity functioning and quality of life in patients who suffer from lower-extremity peripheral artery disease (PAD). We will randomize 106 patients to one of two groups that either receive leg HT or a sham intervention. The primary study outcome is the change in 6-minute walk distance between baseline and the 12-week follow up. Secondary outcomes include changes in the short physical performance battery score, handgrip strength, quality of life (measured by the Walking Impairment Questionnaire and Short-Form (SF)-36 Questionnaire), calf muscle strength (measured using a calf ergometer), size (measured by magnetic resonance imaging) and bioenergetics (assessed using phosphorus-31 magnetic resonance spectroscopy), and physical activity (measured by accelerometer).

DETAILED DESCRIPTION:
The lack of accessible therapies amenable for application in the home setting is a major obstacle for treating patients who suffer from lower-extremity peripheral artery disease (PAD). The investigators will determine whether unsupervised, home-based leg heat therapy (HT) improves walking performance compared to a sham intervention. Leg HT will be applied using water-circulating trousers coupled with a water pump and a water heater. Patients will be randomized into one of two groups: those receiving HT (n=53) or those receiving a sham treatment (n=53).The water heater and pump given to participants in the HT group will be adjusted to circulate water at 42ºC through the trousers. In the sham group, water at 33ºC will be circulated through the trousers. Participants will be asked to apply the therapy daily for 90 min for 3 consecutive months. Outcomes will be assessed at baseline, at the completion of the intervention (end of week 12) and at a follow-up visit, 12 weeks after the end of the intervention (week 24). The primary study outcome is the change in 6-minute walk distance between baseline and the 12-week follow up. Secondary outcomes include changes in the short physical performance battery score, which combines performance in walking speed, standing balance, and repeated chair rises, changes in handgrip strength, perceived quality of life (measured by the Walking Impairment Questionnaire and Short-Form (SF)-36 Questionnaire), calf muscle strength (measured using a calf ergometer), size (measured by magnetic resonance imaging) and bioenergetics (assessed using phosphorus-31 magnetic resonance spectroscopy), and physical activity (measured by accelerometer).

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 50 years
* Resting ankle-brachial index (ABI) of 0.9 or less in at least one leg. Individuals with a resting ABI between 0.91 and 1.00 at baseline will be eligible if their ABI drops by 20% or greater following a heel-rise test.

Exclusion Criteria:

* Critical limb ischemia (ischemic rest pain or ischemia-related, non-healing wounds or tissue loss)
* Prior foot or leg amputation
* Exercise tolerance limited by factors other than leg pain (e.g. angina, arthritis, severe lung disease, etc).
* Recent (<3 months) lower-extremity revascularization or orthopedic surgery
* Use of walking aid other than a cane
* Active cancer
* Chronic kidney disease (eGFR <30 by MDRD or Mayo or Cockcroft-Gault formula)
* Class 2 or 3 obesity (BMI ≥ 35 kg/m2)
* Unable to fit into water-circulating trousers
* A Mini-Mental Status Examination score <23
* Impaired thermal sensation in the leg

As this study involves MR imaging, patients that have contraindications to MRI will be included in the study but will not be allowed to participate in the MRI experiment. Information about biomedical devices that may pose a risk to patients undergoing MRI is available on the Internet at www.MRIsafety.com. These exclusions include: cardiac pacemaker, implanted cardiac defibrillator, aneurysm clips, carotid artery vascular clamp, neurostimulator, insulin or infusion pump, implanted drug infusion device, bone growth/fusion stimulator, cochlear, otologic, or ear implant and history of claustrophobia or who are unable to lie flat or who do not fit inside the bore of the scanner.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk distance | Baseline to 3-month follow-up
  The investigators will determine whether daily leg heat therapy for 90 min using water-circulating trousers perfused with water heated to 42ºC improves the 6-minute walk distance at 3-month follow-up compared to a sham treatment.

SECONDARY OUTCOMES:
Change in Walking Impairment Questionnaire (WIQ) score | Baseline to 3-month follow-up
  This disease-specific questionnaire assess the ability of patients with PAD to walk defined distances and speeds and to climb stairs, with scores ranging from 0 to 100. Higher scores are reflective of better community-based walking ability. The investigators will determine whether leg heat therapy improves the WIQ score at 3-month follow-up compared to the sham treatment.
Change in Short-Form (SF)-36 Questionnaire score | Baseline to 3-month follow-up
  Health-related quality of life (HRQOL) will be assessed using the short-form SF-36 questionnaire, which is composed of 8 subscales. Each subscale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability. The investigators will determine whether leg heat therapy improves the SF-36 score at 3-month follow-up compared to the sham treatment.
Change in Short Physical Performance Battery (SPPB) score | Baseline to 3-month follow-up
  The SPPB combines data from the usual paced 4-m walking velocity, time to rise from a seated position 5 times, and standing balance. The timed results of the subtests will be converted to an ordinal scale ranging from 0 (worst performance) to 12 (best performance). The investigators will determine whether leg heat therapy improves the SPPB score at 3-month follow-up compared to the sham treatment.
Change in handgrip strength | Baseline to 3-month follow-up
  The assessment of maximal handgrip strength will be will performed using a hand dynamometer. The investigators will determine whether leg heat therapy improves handgrip strength at 3-month follow-up compared to the sham treatment.
Change in systolic blood pressure | Baseline to 3-month follow-up
  The systolic blood pressure will be measured in triplicate using a blood pressure monitor. The investigators will determine whether leg heat therapy improves systolic blood pressure at 3-month follow-up compared to the sham treatment.
Change in diastolic blood pressure | Baseline to 3-month follow-up
  The diastolic blood pressure will be measured in triplicate using a blood pressure monitor. The investigators will determine whether leg heat therapy improves blood pressure at 3-month follow-up compared to the sham treatment.
Change in triceps surae volume | Baseline to 3-month follow-up
  The volume of calf muscles will be determined using magnetic resonance (MR) images. The investigators will determine whether leg heat therapy improves calf muscle volume at 3-month follow-up compared to the sham treatment.
Change in triceps surae intramuscular fat content | Baseline to 3-month follow-up
  The intramuscular fat content of calf muscles will be determined using magnetic resonance (MR) images. The investigators will determine whether leg heat therapy reduces intramuscular fat content at 3-month follow-up compared to the sham treatment.
Change in the time constant for phosphocreatine recovery after dynamic exercise | Baseline to 3-month follow-up
  Magnetic resonance spectroscopy tuned to phosphorous (31PMRS) will be used to measure the time constant for PCr recovery (τ) after dynamic planar flexion exercise. The investigators will determine whether leg heat therapy reduces the time constant for PCr recovery at 3-month follow-up compared to the sham treatment.
Change in maximal plantar flexor strength | Baseline to 3-month follow-up
  The maximal voluntary contraction (MVC) strength of the plantar flexor muscles will be assessed using an MR-compatible ergometer (Trispect, Ergospect GmbH, Innsbruck, Austria), Participants will be asked to perform three 4-5 s plantar-flexor MVCs separated by a one-minute rest period. The MVC torque will be considered the highest peak torque value measured over the three trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided